CLINICAL TRIAL: NCT00029874
Title: Minocycline Dosing and Safety in Huntington's Disease
Brief Title: Minocycline in Patients With Huntington's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: FD-R-1968-01
Record Dates: First submitted 2002-01-24; First posted 2002-01-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2004-12

CONDITIONS: Huntington's Disease
Keywords: Tetracyclines; Dose-Response Relationship, Drug
MeSH Terms: conditions — Huntington Disease | interventions — Minocycline

INTERVENTIONS:
Drug: Minocycline

SUMMARY:
This is a study to determine whether treatment with minocycline is safe and tolerable in patients with Huntington's disease (HD) and whether minocycline reduces symptoms of HD in these patients.

DETAILED DESCRIPTION:
Huntington's disease (HD) is a dominantly inherited disorder. It is uniformly progressive and there is no known effective treatment or cure. The pathogenesis is largely unknown; however, recent studies implicate caspase activation, glutamate excitotoxicity, and free radical toxicity as possible causes of HD. Pharmacological agents that block these pathways may be therapeutic in HD. Minocycline is an antibiotic that also inhibits caspase-1 and caspase-3 expression, and inducible nitric oxide synthetase activity, which are factors that may play an important role in the mechanisms of neuropathology in HD.

Two dosages of minocycline or placebo will be given to ambulatory patients with HD over an 8-week period and the tolerability will be compared. Additional measures of safety and the change in motor, behavior, cognitive, and function features will be examined.

ELIGIBILITY:
Inclusion criteria:

* Clinical features of Huntington's disease (HD) and a confirmatory family history of HD and/or a CAG repeat expansion of at least 37
* Stage I, II, or III of illness (TFC greater than or equal to 5)
* Ambulatory and not requiring skilled nursing care
* Patients must use effective birth control
* Concurrent psychotropic medications must be at stable dose for at least 4 weeks prior to study
* WBC count at least 3,800/mm3
* Creatinine no greater than 2.0
* Alanine aminotransferase (ALT) no greater than 2 times upper limit of normal

Exclusion criteria:

* Prior minocycline use within 2 months of baseline visit
* History of known sensitivity or intolerability to minocycline or any other tetracycline
* History of vestibular disease
* Use of any investigational drug within 30 days of baseline visit
* Treatment with any drug that may cause lupus-like symptoms (e.g., procainamide or hydralazine) within 4 weeks of baseline visit
* Pregnant or nursing
* Underlying hematologic, hepatic, or renal disease
* Evidence of unstable medical illness
* Illness that requires use of coumadin
* Unstable psychiatric illness defined as psychosis (hallucinations or delusions), untreated major depression within 90 days of baseline visit, or suicidal ideation
* Substance (alcohol or drug) abuse within 1 year of baseline visit
* History of systemic lupus erythematosis (SLE) or a history of SLE in a first-degree relative
* Positive ANA screening (at or above 1:80)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63
Dates: Start 2001-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States